CLINICAL TRIAL: NCT03768791
Title: Heart Rate Variability in Patients With Failed Back Surgery Syndrome, Treated With Spinal Cord Stimulation
Brief Title: HRV in Patients Treated With Spinal Cord Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moens Maarten (Other)
Responsible Party: Sponsor-Investigator, Moens Maarten, principal investigator, Universitair Ziekenhuis Brussel
Organization: Universitair Ziekenhuis Brussel (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: SYNCHRO
Record Dates: First submitted 2018-11-28; First posted 2018-12-07 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Failed Back Surgery Syndrome
Keywords: Spinal Cord Stimulation; Heart rate variability
MeSH Terms: conditions — Failed Back Surgery Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCS off (Experimental)
  Interventions: Other: SCS is switched off
- SCS on (Experimental)
  Interventions: Other: SCS is switched on

INTERVENTIONS:
Other: SCS is switched off — Spinal cord stimulator is switched off for 12 hours
  Arms: SCS off
Other: SCS is switched on — Spinal cord stimulator is on
  Arms: SCS on

SUMMARY:
This study is an observatory single center study investigating heart rate variability during on and off states of the spinal cord stimulator, in patients with failed back surgery syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years old.
* Diagnosis of FBSS (Failed conservative treatments for pain including but not limited to pharmacological therapy and physical therapy) and currently being treated with spinal cord stimulation.
* Cognitive and language functioning enabling coherent communication between the examiner and the participant.

Exclusion Criteria:

* The presence of one or more coexisting conditions known to affect HRV analysis (including but not limited to atrial fibrillation, numerous atrial or ventricular extra beats, paced rhythm, left ventricular bundle branch block, cancer, kidney or hepatic failure, and diabetes mellitus (autonomic nervous system dysfunction)).
* The use of medication that directly modifies autonomic control (for example beta-blockers).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Heart rate variability changes | Two times on the same day; once while SCS is switched off and once while SCS is switched on. Total study duration lasts one day.
  The investigators will examine the difference in heart rate variability between both measurements (SCS on versus SCS off)

SECONDARY OUTCOMES:
Pain intensity scores | Two times on the same day; once while SCS is switched off and once while SCS is switched on. Total study duration lasts one day.
  Pain intensity scores on a visual analogue scale ranging from zero (no pain) towards 10 (worst possible pain).

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Moens, Prof. dr., Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Jette, Brussels Capital, Belgium

REFERENCES:
- [Background] Kalmar Z, Kovacs N, Balas I, Perlaki G, Plozer E, Orsi G, Altbacker A, Schwarcz A, Hejjel L, Komoly S, Janszky J. Effects of spinal cord stimulation on heart rate variability in patients with chronic pain. Ideggyogy Sz. 2013 Mar 30;66(3-4):102-6. PMID 23750425